CLINICAL TRIAL: NCT00340496
Title: Analysis of NF2 Mutations in Radiation-Related Neural Tumors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996027; OH96-C-N027
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-07

CONDITIONS: Neural Tumors
Keywords: Schwannoma; Meningioma; Follow-Up; Radiation Therapy; Cohort
MeSH Terms: conditions — Neurilemmoma; Meningioma

SUMMARY:
Adults treated with X-rays in childhood for benign conditions such as enlarged tonsils and adenoids have an increased risk of developing nervous system tumors. The risk is highest for schwannomas (RR of 33.1, 95% CI of 9.4-116.5), intermediate for meningiomas (RR of 9.5, 95% CI of 3.5-25.7) and lowest for gliomas (RR of 2.6, 95% CI of 0.8-8.6).

Studies of sporadic tumors of these types have demonstrated the presence of somatic mutations in the NF2 gene. Because these mutations are not usually seen in other types of tumors, they are believed to be what caused the sporadic neural tumors to develop. Germline mutations in the same gene are responsible for the autosomal dominant disorder known as neurofibromatosis 2 (NF2) which is characterized by the development of similar types of neural tumors.

The purpose of the proposed study is to determine if neural tumors that developed in people who were treated with X-rays in childhood also have somatic NF2 mutations. This will be done using DNA from paraffin-embedded neural tumors that developed in ~ 112 individuals treated with X-rays in childhood for benign head and neck conditions. These individuals are from a cohort of over 4,000 irradiated persons followed by Michael Reese Hospital in Chicago since 1974. If we find NF2 mutations in the radiation-related tumors, we will determine whether they are somatic or germline by looking for NF2 mutations in DNA from buccal cells of the patients with the studied tumors. We expect that most patients will have NF2 mutations only in tumor DNA. However, there is a remote possibility that one or more patients may have a germline NF2 mutation and thus an increased risk of developing neural tumors even in the absence of X-ray treatment. We will then compare the types and frequencies of the somatic NF2 mutations with those found in sporadic neural tumors. If we do not find somatic NF2 mutations in the radiation-related tumors, we will conclude that X-rays caused neural tumors to develop through interactions with another gene or genes. Either result will contribute to our knowledge of radiation tumorigenesis.

We will send letters describing this study to patients from the Michael Reese Hospital cohort who have developed radiation-related neural tumors. Those who consent to take part in it will be asked for permission to obtain paraffin blocks from any neural tumor that they have had removed and to donate buccal cells for NF2 mutation studies. Finally, they will also be asked to complete a questionnaire that will help us update their medical history and obtain a medical history on close blood relatives.

DETAILED DESCRIPTION:
Adults treated with X-rays in childhood for benign conditions such as enlarged tonsils and adenoids have an increased risk of developing nervous system tumors. The risk is highest for schwannomas (RR of 33.1, 95% CI of 9.4-116.5), intermediate for meningiomas (RR of 9.5, 95% CI of 3.5-25.7) and lowest for gliomas (RR of 2.6, 95% CI of 0.8-8.6).

Studies of sporadic tumors of these types have demonstrated the presence of somatic mutations in the NF2 gene. Because these mutations are not usually seen in other types of tumors, they are believed to be what caused the sporadic neural tumors to develop. Germline mutations in the same gene are responsible for the autosomal dominant disorder known as neurofibromatosis 2 (NF2) which is characterized by the development of similar types of neural tumors.

The purpose of the proposed study is to determine if neural tumors that developed in people who were treated with X-rays in childhood also have somatic NF2 mutations. This will be done using DNA from paraffin-embedded neural tumors that developed in ~ 112 individuals treated with X-rays in childhood for benign head and neck conditions. These individuals are from a cohort of over 4,000 irradiated persons followed by Michael Reese Hospital in Chicago since 1974. If we find NF2 mutations in the radiation-related tumors, we will determine whether they are somatic or germline by looking for NF2 mutations in DNA from buccal cells of the patients with the studied tumors. We expect that most patients will have NF2 mutations only in tumor DNA. However, there is a remote possibility that one or more patients may have a germline NF2 mutation and thus an increased risk of developing neural tumors even in the absence of X-ray treatment. We will then compare the types and frequencies of the somatic NF2 mutations with those found in sporadic neural tumors. If we do not find somatic NF2 mutations in the radiation-related tumors, we will conclude that X-rays caused neural tumors to develop through interactions with another gene or genes. Either result will contribute to our knowledge of radiation tumorigenesis.

We will send letters describing this study to patients from the Michael Reese Hospital cohort who have developed radiation-related neural tumors. Those who consent to take part in it will be asked for permission to obtain paraffin blocks from any neural tumor that they have had removed and to donate buccal cells for NF2 mutation studies. Finally, they will also be asked to complete a questionnaire that will help us update their medical history and obtain a medical history on close blood relatives.

ELIGIBILITY:
* INCLUSION CRITERIA:

Members of a cohort of 4,296 patients who received conventional (200 kV) radiation treatment to the head and neck for benign conditions before their 16th birthday.

All of the patients were treated at Michael Reese Hospital, Chicago, between 1939 and 1962.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112
Dates: Start 1996-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States